CLINICAL TRIAL: NCT00697060
Title: A Multicenter, Phase II Trial of the Safety and Efficacy of Amplimexon® (Imexon for Injection) in Combination With Taxotere® (Docetaxel) for Previously Treated Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Safety and Efficacy Trial of Amplimexon Plus Taxotere in Metastatic Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study cancelled prior to start due to change in company priorities.
Sponsor: AmpliMed Corporation (Industry)
Responsible Party: Evan Hersh, AmpliMed
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP024
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Metastatic; Previously treated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one; Docetaxel

ARMS (1):
- Stage 1/2 (Experimental): Imexon plus docetaxel
  Interventions: Drug: Imexon + docetaxel

INTERVENTIONS:
Drug: Imexon + docetaxel — Imexon at 1300 mg/m2 days 1-5 Docetaxel at 75 mg/m2 day 1
  Other Names: Amplimexon; Taxotere

SUMMARY:
Protocol AMP-024 is a Phase 2 study of imexon plus docetaxel for patients with previously treated lung cancer that has spread in the body. Docetaxel is approved by the Food and Drug Administration (FDA) as a second line therapy for this cancer. The imexon is administered on days 1-5 and the docetaxel on day 1 of every 3 week cycle. The objective of the protocol is to determine if the combination of imexon plus docetaxel is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically or cytologically confirmed NSCLC.
2. Subject with metastatic disease (Appendix D) who have received no more than 2 prior chemotherapy regimens for their metastatic disease.

   * Adjuvant chemotherapy is considered one prior regimen.
   * Immunological and targeted agents such as bevacizumab, erlotinib or gefitinib are considered prior regimens.
3. Subjects must have at least one measurable lesion by RECIST criteria (Appendix C). If the only measurable lesion is a lymph node, it must measure at least 20 mm in LD, and if the only target lesion is a single lesion, a cytological or histological confirmation of NSCLC is required.
4. Resolution of all chemotherapy or radiotherapy-related toxicities to CTCAE grade 1 or lower, except for stable sensory neuropathy of < grade 2 and/or alopecia.
5. Men and women age > 18 years.
6. ECOG performance status of 0 - 1 (Appendix E).
7. Not pregnant nor lactating.
8. If of child bearing potential must be able and agree to use adequate contraception.
9. Adequate renal function defined by:

   * serum creatinine level < 2.0 mg/dL.
10. G6PD (quantitative) greater than or equal to the lower limit of normal.
11. Adequate hematologic function defined by:

    * absolute neutrophil count (ANC) >1,500/mm³, and
    * platelet count > 100,000/mm³, and
    * hemoglobin level > 9 g/dL.
12. Adequate hepatic function defined by:

    * total bilirubin level < ULN, and
    * AST and ALT levels < 1.5 x ULN
    * Alkaline phosphatase < 2.5x ULN
13. Prior brain metastasis are allowed but must have been treated and controlled for > 1 month prior and be off steroids.
14. Subjects willing and able to comply with the study protocol for the duration of the study.
15. Able to render written informed consent and to follow protocol requirements.

Exclusion Criteria:

1. Subjects who have received previous treatment with docetaxel.
2. Subjects who have received chemotherapy or radiation treatments within 4 weeks of study treatment start.
3. Prior high dose chemotherapy with hematopoietic stem cell rescue within the past two years.
4. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen and/or the medical management of recurrent pleural effusions.
5. Subjects with meningeal carcinomatosis.
6. Women who are pregnant or breast-feeding, women of child bearing potential (WOCBP) with either a positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) or no pregnancy test; WOCBP unless (1) surgically sterile (hysterectomy, or bilateral oophorectomy) or (2) not using adequate measures of contraception in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
7. Severe or uncontrolled intercurrent infection or other illness.
8. Significant cardiovascular disease including but not limited to a history of congestive heart failure of > NYHA grade II (Appendix E), unstable angina or a myocardial infarction within the past six months, or serious and uncontrolled arrhythmia.
9. Subjects with organ allografts.
10. Subjects who have had a prior malignancy, other than carcinoma in situ of the cervix, non-melanoma skin cancer, and superficial bladder cancer unless the prior malignancy was diagnosed and definitively treated > 5 years previously with no subsequent evidence of recurrence.
11. Subjects with pre-existing neuropathy > CTCAE Grade 2.
12. Subjects with other significant disease or disorders that, in the opinion of the Investigator, would exclude the subject from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rates (CR + PR) in subjects with measurable disease will be determined by RECIST methodology. | every 6 weeks

SECONDARY OUTCOMES:
Progression-free survival (PFS), as measured from the date of registration to the date of recorded disease progression (PD) or death from any cause. | throughout the study
Overall survival, as measured from the date of registration to the date of death from any cause. | throughout the study
Stable disease rate at 2 months. | 2 months
Survival at 1-year. | 1 year
Duration of response and stable disease. | throughout the study
Safety parameters (AEs, laboratory parameters, concomitant medication, study drug exposure, drug related toxicities, etc.) | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Evan Hersh, MD, Study Director — AmpliMed Corporation
Locations (3):
- United States (3):
  - USC Norris Cotton Cancer Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mary Crowley Research Center, Dallas, Texas